CLINICAL TRIAL: NCT05614661
Title: Postpartum Intervention for Mothers With Opioid Use Disorders - Brain-Behavior Mechanisms
Brief Title: Postpartum Intervention for Mothers With Opioid Use Disorders
Acronym: PIMO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, James Edward Swain, Associate Professor, Stony Brook University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB2022-00166
Record Dates: First submitted 2022-11-05; First posted 2022-11-14 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Opioid Use Disorder
Keywords: parenting intervention; Opioid Use Disorder; parental stress; maternal brain; evoked response potentials
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: This is a 2-group (Mom Power (MP) vs. control), pre-post RCT of mothers with OUD to test the effect of MP on drug craving, mood and electrophysiological responses to own infant faces (MP n=40; control n= 10)
Masking Description: -it's impossible to mask whether receiving the therapy treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mom Power (Experimental): Mom Power is an evidence-based 13-session psychosocial mother-child group intervention that improves sensitive caregiving, parental stress, and depression
  Interventions: Behavioral: Mom Power
- Control (Sham Comparator): Controls participants for the intervention receive 10 weekly mailings, with content relevant for the postpartum period (i.e., information on baby sleep, developmental milestones, box breathing and other self-care/coping strategies, fun games to play with a baby, and community resources, and general parenting); plus 10 brief check-in phone calls verifying that material was received, and additional longer phone calls to assess any imminent family needs and provide resources as needed/requested.
  Interventions: Behavioral: Mom Power

INTERVENTIONS:
Behavioral: Mom Power — Experimental participants will receive virtual Mom Power via phone/internet connection. Control participants will receive mail information and confirmation phone calls.

SUMMARY:
Opioid use disorder (OUD) is a fast-growing and devastating epidemic in the US with many mothers suffering cravings, depression, impaired interpersonal interactions and maladaptive parenting behaviors that may lead to child maltreatment and costly utilization of foster care. This interdisciplinary multisite project will begin with the high risk R61 phase, in which the investigators will administer the parenting intervention "Mom Power" to mothers with OUD during the first 6 months postpartum and look for effects on drug use, mood and brain mechanisms; and, If validated, the investigators will continue in the R33 with more brain mechanism investigation and outcome studies a larger sample. The completion of this grant will clarify the effects of parenting intervention for mothers with OUD, and yield brain-based biomarkers that may be connected with inexpensive measures toward improved treatment of families suffering OUD, their children and society - which ultimately bears much of the cost for the common trans-generational problems of peripartum drug use.

DETAILED DESCRIPTION:
Postpartum Intervention for Mothers with Opioid Use Disorders - Brain-Behavior Mechanisms Opioid use disorder (OUD) is a fast-growing and devastating epidemic in the US with many suffering comorbid mood disorders. Despite receiving "gold standard" buprenorphine treatment to reduce withdrawal, OUD mothers still suffer have cravings, depression, impaired interpersonal interactions and maladaptive parenting behaviors that may lead to child maltreatment and costly utilization of foster care. Parenting interventions have been established to improve parent mood and sensitive caregiving behaviors for high-risk non-OUD populations. "Mom Power" (MP) is an evidence-based 13-session psychosocial mother-child intervention established to enhance emotionally sensitive caregiving, while concurrently reducing parental stress and depression for non-OUD mothers. The investigators have demonstrated feasibility of with virtual MP (vMP) and for MP with substance use disorders. However, vMP for mothers with OUD has not been studied with respect to drug use reduction or mood improvement. The investigators have also established brain mechanisms that regulate parenting. Recent work from the investigators has established that a parenting intervention for non-OUD mothers was associated with a larger enhancement of evoke potential responses (ERPs) for emotional faces relative to neutral faces and that the magnitude of ERP responses to emotional faces was associated with observed maternal sensitivity. Using functional magnetic resonance imaging (fMRI) of the brain, the investigators have also established a Maternal Behavior Neurocircuit (MBN) that regulates flexible responses to the demands of their own infant - such as to the unique, ethologically salient own-baby cry and face stimuli during the early postpartum period. The investigators have established fMRI maternal brain changes associated with MP in non-OUD mothers, and brain effects of OUD on mothers. However, it is unknown how parental brain mechanisms through which parenting interventions may work for mothers with OUD, such as affecting ERP or fMRI responses to baby stimuli in the MBN. Central hypotheses: Mothers with OUD who get virtual MP (vMP), compared to matched controls, will show improved drug craving, mood, and stress symptoms, via changes in pre-specified MBN brain regions. In the high-risk R61 phase, the investigators will establish if vMP (n=25) for OUD can be implemented and improve mood, reduce drug use and affect ERP brain responses to baby pictures compared with control (n=25). If hypotheses in the R61 are confirmed, the investigators will confirm and expand this breakthrough with the R33 Phase (n=160, 80/group), adding richer maternal outcome measures and MBN fMRI. This research will elucidate the effects of parenting intervention MP on drug use and brain function for OUD mothers - with translational potential for biomarker and treatment development.

ELIGIBILITY:
Inclusion Criteria:

* mothers aged 18-50 from SBU or UM with diagnosis of Opioid Use Disorder (OUD); and/or receiving medication assisted treatment (such as buprenorphine or methadone)
* with a child aged 5 or less
* able to read, hear and understand English adequately enough to provide informed consent

Exclusion Criteria:

1. require immediate clinical care for suicidal/homicidal risk or psychosis (please see Protection of Human Subjects section for clinical management of suicidal risk);
2. For magnetic resonance imaging (MRI) of the brain, potential participants will be excluded if they:

1) have ferromagnetic metal in their heads 2) have severe claustrophobia that prevents participation in the neuroimaging 3) have serious neurological condition that could interfere with neuroimaging, including a brain tumor, multiple sclerosis or significant head trauma 4) Exclusion from MRI does not necessarily exclude participant from study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Mom Power for mothers
Enrollment: 50 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
R61 Milestone 1 | <2 years
  To recruit at least N = 50 participants in 11.25 months for the expanded number in the R33
R61 Milestone 2 | <2 years
  To end with 80% of mothers in the MP condition attending >=80% of sessions
R61 Milestone 3 | <2 years
  To end with >=70% yielding satisfactory pre- and post-intervention ERP and fMRI data
R61 Milestone 4 | <2 years
  To show that vMP for OUD significantly affects ERP (LPP and N170) and drug craving, mood, and parenting stress (P<0.05)

CONTACTS AND LOCATIONS:
Overall Officials: James E Swain, MD, PhD, Principal Investigator — Stony Brook University
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Stony Brook University, Stony Brook, New York

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Rosenblum K, Lawler J, Alfafara E, Miller N, Schuster M, Muzik M. Improving Maternal Representations in High-Risk Mothers: A Randomized, Controlled Trial of the Mom Power Parenting Intervention. Child Psychiatry Hum Dev. 2018 Jun;49(3):372-384. doi: 10.1007/s10578-017-0757-5. PMID 28936602
- [Background] Muzik M, Rosenblum KL, Alfafara EA, Schuster MM, Miller NM, Waddell RM, Stanton Kohler E. Mom Power: preliminary outcomes of a group intervention to improve mental health and parenting among high-risk mothers. Arch Womens Ment Health. 2015 Jun;18(3):507-21. doi: 10.1007/s00737-014-0490-z. Epub 2015 Jan 11. PMID 25577336
- [Background] Ho SS, Muzik M, Rosenblum KL, Morelen D, Nakamura Y, Swain JE. Potential Neural Mediators of Mom Power Parenting Intervention Effects on Maternal Intersubjectivity and Stress Resilience. Front Psychiatry. 2020 Dec 8;11:568824. doi: 10.3389/fpsyt.2020.568824. eCollection 2020. PMID 33363481
- [Background] Swain JE, Ho SS, Rosenblum KL, Morelen D, Dayton CJ, Muzik M. Parent-child intervention decreases stress and increases maternal brain activity and connectivity during own baby-cry: An exploratory study. Dev Psychopathol. 2017 May;29(2):535-553. doi: 10.1017/S0954579417000165. PMID 28401845
- [Background] Swain JE, Ho SS, Fox H, Garry D, Brummelte S. Effects of opioids on the parental brain in health and disease. Front Neuroendocrinol. 2019 Jul;54:100766. doi: 10.1016/j.yfrne.2019.100766. Epub 2019 May 22. PMID 31128130
- [Background] Swain JE, Ho SS. Early postpartum resting-state functional connectivity for mothers receiving buprenorphine treatment for opioid use disorder: A pilot study. J Neuroendocrinol. 2019 Sep;31(9):e12770. doi: 10.1111/jne.12770. Epub 2019 Jul 29. PMID 31287922
- [Background] Swain JE, Ho SS. Opioids and maternal brain-behavior adaptation. Neuropsychopharmacology. 2021 Jan;46(1):265-266. doi: 10.1038/s41386-020-00858-7. No abstract available. PMID 32913343
- [Background] Swain JE, Ho SS. Reduced Child-Oriented Face Mirroring Brain Responses in Mothers With Opioid Use Disorder: An Exploratory Study. Front Psychol. 2022 Feb 4;12:770093. doi: 10.3389/fpsyg.2021.770093. eCollection 2021. PMID 35185679
- [Background] Swain JE, Ho SS. Brain circuits for maternal sensitivity and pain involving anterior cingulate cortex among mothers receiving buprenorphine treatment for opioid use disorder. J Neuroendocrinol. 2023 Jul;35(7):e13316. doi: 10.1111/jne.13316. Epub 2023 Jul 25. PMID 37491982
- [Background] Ho SS, Nakamura Y, Gopang M, Swain JE. Intersubjectivity as an antidote to stress: Using dyadic active inference model of intersubjectivity to predict the efficacy of parenting interventions in reducing stress-through the lens of dependent origination in Buddhist Madhyamaka philosophy. Front Psychol. 2022 Jul 29;13:806755. doi: 10.3389/fpsyg.2022.806755. eCollection 2022. PMID 35967689